CLINICAL TRIAL: NCT02362022
Title: Comparison of Two Different Doses of Intravenous Morphine on Desflurane Consumption and Recovery Time in Patients Undergoing Total Abdominal Hysterectomy
Brief Title: The Effects of Morphine on Desflurane Consumption and Recovery Time
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, CAGLA BALI,MD, medical doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14.09.2007/88-4
Record Dates: First submitted 2015-02-04; First posted 2015-02-12 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-06

CONDITIONS: Abdominal Hysterectomy (& Wertheim)
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Saline (Placebo Comparator): Group Saline (Group S) received i.v saline 0.9 % in 10 ml volume (n=30)
  Interventions: Drug: Morphine
- Group Morphine 1 (Active Comparator): Group Morphine 1 (Group M1) received i.v morphine 0.1 mg kg-1, in 10 ml volume (n=30)
  Interventions: Drug: Morphine
- Group Morphine 2 (Active Comparator): Group Morphine 2 (Group M2) received i.v morphine 0.2 mg kg-1, in 10 ml volume (n=30)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Group Saline (Group S): Received i.v saline 0.9 % in 10 ml volume (n=30) Group Morphine 1 (Group M1): Received i.v morphine 0.1 mg kg-1 in 10 ml volume (n=30) Group Morphine 2 (Group M2): Received i.v morphine 0.2 mg kg-1 in 10 ml volume (n=30)

SUMMARY:
Combination of volatile and opioid agents are used to achieve unconsciousness, haemodynamic stability and analgesia for surgical prosedures. This prospective, randomized, double-blind, controlled study evaluates the effects of two different doses of morphine sulphate (0.1 mg/kg and 0.2 mg/kg), on desflurane consumption, recovery characteristics, postoperative analgesic requirements and side effects during total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* undergoing total abdominal hysterectomy with general anaesthesia

Exclusion Criteria:

* renal dysfunction (cre>1.2), liver failure, cardiovascular, psychiatric, allergic and metabolic disorders

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
postoperative desflurane consumption | postoperative first hour
sedation scores for OASS scale | postoperative first hour

CONTACTS AND LOCATIONS:
Overall Officials: cagla bali, Principal Investigator — Baskent University
Locations (1):
- Baskent University School of Medicine Adana Teaching and Research Hospital, Adana, Turkey (Türkiye)